CLINICAL TRIAL: NCT01468974
Title: A Clinical Evaluation of the Abbott Vascular ESPRIT BVS (Bioresorbable Vascular Scaffold) System for the Treatment of Subjects With Symptomatic Claudication From Occlusive Vascular Disease of the Superficial Femoral (SFA) or Common or External Iliac Arteries.
Brief Title: ESPRIT I: A Clinical Evaluation of the Abbott Vascular ESPRIT BVS (Bioresorbable Vascular Scaffold) System
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Abbott Medical Devices (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 11-113
Record Dates: First submitted 2011-11-02; First posted 2011-11-10 (Estimated); Results first posted 2019-02-04 (Actual); Last update posted 2019-02-04 (Actual); Status verified 2018-02

CONDITIONS: Atherosclerosis; Peripheral Vascular Disease; Claudication
MeSH Terms: conditions — Atherosclerosis; Peripheral Vascular Diseases; Intermittent Claudication

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- ESPRIT BVS (Other): Subjects receiving the ESPRIT BVS for the treatment of symptomatic claudication from occlusive vascular disease of the superficial femoral (SFA) or common or external iliac arteries.
  Interventions: Device: ESPRIT BVS

INTERVENTIONS:
Device: ESPRIT BVS — Subjects receiving ESPRIT BVS for the treatment of symptomatic claudication from occlusive vascular disease of the superficial femoral (SFA) or common or external iliac arteries

SUMMARY:
The purpose of the ESPRIT I Clinical Investigation is to evaluate the safety and performance of the ESPRIT BVS in subjects with symptomatic claudication from occlusive vascular disease of the superficial femoral (SFA) or common or external iliac arteries.

ELIGIBILITY:
Inclusion Criteria:

1. Subject is ≥ 18 and ≤ 80 years of age at the time of signing informed consent.
2. Subject is diagnosed as having symptomatic claudication (Rutherford-Becker Clinical Category 1-3).

   For subjects with bilateral lesions, the higher Rutherford-Becker Clinical Category limb will be considered the target extremity to be treated in this trial.

   If both limbs are of the same Rutherford Becker Clinical Category, the target extremity will be selected based on investigator discretion.
3. Subject or legally authorized representative has been informed of the nature of the study, agrees to its provisions, and is able to provide informed consent.
4. Subject agrees to undergo all protocol-required follow-up examinations and requirements at the investigational site.
5. Female subject of childbearing potential must: have had a negative pregnancy test within 14 days before treatment; not be nursing at the time of the study procedure and agree at time of consent to use birth control during participation in this trial.
6. Subject has life expectancy > 12 months.
7. Subject is able to take clopidogrel or prasugrel (or ticlopidine, if the subject cannot take clopidogrel or prasugrel) and acetylsalicylic acid (aspirin).
8. Subject must agree not to participate in any other clinical investigation for a period of 12 months following the index procedure. This includes clinical trials of medications and invasive procedures. Questionnaire-based studies, or other studies that are non-invasive and do not require medication are allowed.

Angiographic Inclusion Criteria

1. A single de novo native disease segment of the superficial femoral (SFA) or common or external iliac arteries of the target extremity located within the following anatomical parameters:

   Iliac
   * Proximal margin of target lesion is ≥ 2.5 cm distal to the aortic bifurcation in common iliac artery
   * Distal margin of target lesion is ≥ 1.5 cm proximal to the location of inguinal ligament

   SFA
   * Proximal margin of target lesion is ≥ 1 cm distal to the common femoral artery bifurcation
   * Distal margin of target lesion is ≤ 25 cm distal to the common femoral artery bifurcation
2. Vessel diameter from ≥ 5.5 mm to ≤ 6.5 mm evaluated by on-line quantitative vascular angiography (QVA) after pre-dilatation per core laboratory guidelines
3. Target lesion is ≥ 50% DS
4. Target lesion length ≤ 50 mm
5. Patent inflow artery free from significant lesion (≥ 50% DS and < 100% DS) as confirmed by angiography (treatment of the target lesion acceptable after successful treatment of inflow artery lesion)
6. Patent popliteal artery free from significant lesion (≥ 50% DS) with at least one patent distal outflow artery (anterior tibial, posterior tibial, or peroneal) that provides in-line circulation to the lower leg and foot, as confirmed by angiography

Exclusion Criteria:

1. A platelet count <100,000 cells/mm3 or >700,000 cells/mm3; a white blood cell count (WBC) <3,000 cells/mm3; or hemoglobin < 10.0 g/dL
2. Acute or chronic renal dysfunction (creatinine > 2.5 mg/dl or >176μmol/L)
3. Severe liver impairment as defined by total bilirubin ≥ 3 mg/dl or two times increase over the normal level of serum glutamic oxaloacetic transaminase (SGOT) or serum glutamic pyruvic transaminase (SGPT).
4. Known allergies to the following: aspirin, clopidogrel, prasugrel or ticlopidine, heparin, contrast agent (that cannot be adequately premedicated), or drugs similar to everolimus (i.e. tacrolimus, sirolimus, zotarolimus) or other macrolides.
5. Subject requires planned procedure that would necessitate the discontinuation of clopidogrel, prasugrel or ticlopidine.
6. Subject has had or will require treatment with drug eluting stent (DES) or drug coated balloon (DCB) within 6 months pre- or post-index procedure.
7. Subject is unable to walk.
8. Subject has undergone any non-iliac percutaneous intervention, e.g. coronary, carotid, < 30 days prior to the planned index procedure.
9. Subject has received, or is on the waiting list for, a organ transplant.
10. Subject is on chronic hemodialysis.
11. Subject has uncontrolled diabetes mellitus (DM) (HbA1c ≥ 7.0%).
12. Subject has had a myocardial infarction (MI) within the previous 30 days of the planned index procedure.
13. Subject has had a stroke within the previous 30 days of the planned index procedure and/or has deficits from a prior stroke that limits the subject's ability to walk.
14. Subject has unstable angina defined as rest angina with ECG changes.
15. Subject has a groin infection, or an acute systemic infection that has not been treated successfully or is currently under treatment.
16. Subject has acute thrombophlebitis or deep vein thrombosis in either extremity.
17. Subject has other medical illnesses (e.g., cancer or congestive heart failure) that may cause the subject to be non-compliant with protocol requirements, confound the data interpretation or is associated with limited life-expectancy, i.e., less than 12 months.
18. Subject is currently participating in an investigational drug, biologic, or device study that has not completed the primary endpoint or that clinically interferes with the current study endpoints. (Note: Trials requiring extended follow-up for products that were investigational, but have since become commercially available, are not considered investigational trials.)
19. Subject is unable to understand or unwilling to cooperate with study procedures.
20. Subject requires general anesthesia for the procedure.
21. Subject has ischemic or neuropathic ulcers on either foot.
22. Subject has prior minor or major amputation of either lower extremity.
23. Subject is part of a vulnerable population who, in the judgment of the investigator, is unable to give informed consent for reasons of incapacity, immaturity, adverse personal circumstances or lack of autonomy. This may include: Individuals with mental disability, persons in nursing homes, children, impoverished persons, subjects in emergency situations, homeless persons, nomads, refugees, and those incapable of giving informed consent. Vulnerable populations also may include members of a group with a hierarchical structure such as university students, subordinate hospital and laboratory personnel, employees of the sponsor, members of the armed forces, and persons kept in detention.

Angiographic Exclusion Criteria

1. Contralateral lesion distal to the location of inguinal ligament that requires treatment within 30 days before or after the procedure. (Contralateral iliac artery lesions may be treated during the procedure if necessary for contralateral approach to the target lesion).
2. Target extremity has an angiographically significant (> 50% DS) lesion located distal to the target lesion.
3. Acute ischemia of the target extremity
4. Target extremity has been previously treated with any of the following: surgical bypass or endarterectomy.
5. Target vessel has been previously treated with any of the following: stent, laser, atherectomy, surgical bypass, or endarterectomy.
6. Total occlusion (100% DS) of the ipsilateral inflow artery.
7. Angiographic evidence of thrombus in target vessel.
8. The target lesion requires treatment with a device other than percutaneous transluminal angioplasty (PTA) (e.g. but not limited to, directional atherectomy, excimer laser, rotational atherectomy, brachytherapy, cryoplasty, etc.)
9. Target lesion is within or adjacent to an aneurysm.
10. Subject has angiographic evidence of thromboembolism or atheroembolism from treatment of an ipsilateral iliac lesion, or from crossing or pre-dilating the target lesion.
11. Target lesion has moderate-to-severe calcification with either of the following characteristics:

    * Circumferential orientation
    * Thickness > 2 mm in either radial or longitudinal direction
12. Subject has an abdominal aortic aneurysm > 3 cm or history of aortic revascularization.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2011-11; Primary Completion 2015-08 (Actual); Study Completion 2015-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Johannes Lammer, Prof. Dr., Principal Investigator — Medical University of Vienna
Locations (8):
- Medical University of Vienna, Vienna, Austria
- Belgium (4):
  - Abbott Vascular International BVBA, Brussels
  - Sint-Blasius Hospital, Dendermonde
  - Oost Limburg Ziekenhuis, Genk
  - Gent University Hospital, Ghent
- Clinique Pasteur, Toulouse, France
- Germany (2):
  - Herzzentrum Bad Krozingen, Bad Krozingen
  - Park-Krankenhaus Leipzig, Leipzig

REFERENCES:
- [Derived] Lammer J, Bosiers M, Deloose K, Schmidt A, Zeller T, Wolf F, Lansink W, Sauguet A, Vermassen F, Lauwers G, Scheinert D, Popma JJ, McGreevy R, Rapoza R, Schwartz LB, Jaff MR. Bioresorbable Everolimus-Eluting Vascular Scaffold for Patients With Peripheral Artery Disease (ESPRIT I): 2-Year Clinical and Imaging Results. JACC Cardiovasc Interv. 2016 Jun 13;9(11):1178-87. doi: 10.1016/j.jcin.2016.02.051. PMID 27282601

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 35 subjects registered in this study were implanted with the ESPRIT BVS at 7 centers in 4 countries (Belgium, France, Germany and Austria) across Europe. First subject was registered in the ESPRIT I Clinical Investigation on December 20, 2011. The last subject was registered on August 28, 2012.
Period: 1 Month Follow-up
Arm/Group | ESPRIT BVS
Started | 35 (Intent-to-treat (ITT) population)
Completed | 34
Not Completed | 1
Period: 6 Months Follow-up
Arm/Group | ESPRIT BVS
Started | 34
Completed | 34
Not Completed | 0
Period: 1 Year Follow-up
Arm/Group | ESPRIT BVS
Started | 34
Completed | 34
Not Completed | 0
Period: 2 Years Follow-up
Arm/Group | ESPRIT BVS
Started | 34
Completed | 32
Not Completed | 2
Period: 3 Years Follow-up
Arm/Group | ESPRIT BVS
Started | 32
Completed | 26
Not Completed | 6

BASELINE CHARACTERISTICS:
Arm/Group | ESPRIT BVS
Number analyzed (Participants) | 35
Age, Continuous [Mean (Standard Deviation); unit: years] | 65.3 (8.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8
  Male | 27
Region of Enrollment [Number; unit: participants]
  Austria | 4
  Belgium | 20
  France | 3
  Germany | 8

OUTCOME MEASURES:

1. Primary Outcome: Device Success
Description: Study device success is defined on a per device basis, the achievement of successful delivery and deployment of the study device(s) at the intended target lesion and successful withdrawal of the delivery catheter.
Time Frame: On Day 0 (From start of index procedure to end of index procedure)
Population: Intent-to-treat (ITT) population.
Measure: Number; unit: percentage of devices
Arm/Group | ESPRIT BVS
Number analyzed (Participants) | 35
percentage of devices | 100.0

2. Primary Outcome: Technical Success
Description: Technical success is defined on a per lesion basis, the attainment of a final residual stenosis of < 30% at the intended target lesion(s). Standard pre-dilation catheters and post-dilatation catheters (if applicable) may be used. Bailout patients will be included as technical success only if the above criteria are met.
Time Frame: On Day 0 (From start of index procedure to end of index procedure)
Population: ITT population.
Measure: Number; unit: percentage of target lesions
Arm/Group | ESPRIT BVS
Number analyzed (Participants) | 35
percentage of target lesions | 97.1

3. Primary Outcome: Clinical Success
Description: Defined on a per subject basis, as the attainment of a final residual stenosis of < 30% using the study device(s) and/or any adjunctive device at all intended target lesion(s) without complications* within 2 days after the index procedure or at hospital discharge, whichever is sooner. (Note that in the ESPRIT I study, only a single target lesion per subject is permitted to be treated).
  *Includes the following: Death; Amputation; Scaffold Thrombosis; Target Lesion Revascularization (by any percutaneous or surgical means); Target Vessel Revascularization (by any percutaneous or surgical means).
Time Frame: > or = 2 days after the index procedure
Population: ITT population.
Measure: Number; unit: percentage of participants
Arm/Group | ESPRIT BVS
Number analyzed (Participants) | 35
percentage of participants | 97.1

4. Secondary Outcome: Number of Participants With Death
Description: Cardiac death is defined as any death in which a cardiac cause cannot be excluded. (This includes but is not limited to acute myocardial infarction, cardiac perforation/pericardial tamponade, arrhythmia or conduction abnormality,cerebrovascular accident within 30 days of the procedure or cerebrovascular accident suspected of being related to the procedure, death due to complication of the procedure, including bleeding, vascular repair, transfusion reaction, or bypass surgery.)
  -Non-cardiac death is defined as a death not due to cardiac causes (as defined above).
Time Frame: 1 month
Population: ITT population. The number of participants analyzed includes subjects who had available follow up data at that time frame. The number of participants analyzed includes subjects who had available follow up data at that time frame.
Measure: Count of Participants; unit: Participants
Arm/Group | ESPRIT BVS
Number analyzed (Participants) | 35
Participants | 0

5. Secondary Outcome: Number of Participants With Death
Description: as for outcome 4
Time Frame: 6 months
Population: ITT population. Per-subject basis analysis. The number of participants analyzed includes subjects who had available follow up data at that time frame. The analysis population excluded subjects who had lost-to-follow up at that time frame.
Measure: Count of Participants; unit: Participants
Arm/Group | ESPRIT BVS
Number analyzed (Participants) | 34
Participants | 0

6. Secondary Outcome: Number of Participants With Death
Description: as for outcome 4
Time Frame: 1 year
Population: as for outcome 5
Measure: Count of Participants; unit: Participants
Arm/Group | ESPRIT BVS
Number analyzed (Participants) | 34
Participants | 0

7. Secondary Outcome: Number of Participants With Death
Description: as for outcome 4
Time Frame: 2 years
Population: as for outcome 5
Measure: Count of Participants; unit: Participants
Arm/Group | ESPRIT BVS
Number analyzed (Participants) | 33
Participants | 1

8. Secondary Outcome: Number of Participants With Death
Description: as for outcome 4
Time Frame: 3 years
Population: as for outcome 5
Measure: Count of Participants; unit: Participants
Arm/Group | ESPRIT BVS
Number analyzed (Participants) | 29
Participants | 1

9. Secondary Outcome: Number of Participants With Any Amputation of Treated Limb (Minor and Major)
Description: The removal of a body extremity by surgery. For this study, the definition of amputation will only apply to amputations of the limb that was treated.
  A minor amputation will be defined as below-the-ankle; and a major amputation will be defined as limb loss at or proximal to the transtibial level. Major amputations will be specified as below-the-knee and above-the-knee amputations.
Time Frame: 1 month
Population: ITT population. The number of participants analyzed includes subjects who had available follow up data at that time frame.
Measure: Count of Participants; unit: Participants
Arm/Group | ESPRIT BVS
Number analyzed (Participants) | 35
Participants | 0

10. Secondary Outcome: Number of Participants With Any Amputation of Treated Limb (Minor and Major)
Description: as for outcome 9
Time Frame: 6 months
Population: ITT population. The number of participants analyzed includes subjects who had available follow up data at that time frame. The analysis population excluded subjects who had lost-to-follow up at that time frame.
Measure: Count of Participants; unit: Participants
Arm/Group | ESPRIT BVS
Number analyzed (Participants) | 34
Participants | 0

11. Secondary Outcome: Number of Participants With Any Amputation of Treated Limb (Minor and Major)
Description: as for outcome 9
Time Frame: 1 year
Population: as for outcome 10
Measure: Count of Participants; unit: Participants
Arm/Group | ESPRIT BVS
Number analyzed (Participants) | 34
Participants | 0

12. Secondary Outcome: Number of Participants With Any Amputation of Treated Limb (Minor and Major)
Description: as for outcome 9
Time Frame: 2 years
Population: as for outcome 10
Measure: Count of Participants; unit: Participants
Arm/Group | ESPRIT BVS
Number analyzed (Participants) | 33
Participants | 0

13. Secondary Outcome: Number of Participants With Any Amputation of Treated Limb (Minor and Major)
Description: as for outcome 9
Time Frame: 3 years
Population: ITT population. The analysis population excluded subjects who had lost-to-follow up at that time frame.
Measure: Count of Participants; unit: Participants
Arm/Group | ESPRIT BVS
Number analyzed (Participants) | 29
Participants | 0

14. Secondary Outcome: Number of Participants With Limb Salvage (Freedom From Ipsilateral Major Amputations) of the Target Extremity
Description: Amputation:
  The removal of a body extremity by surgery. For this study, the definition of amputation will only apply to amputations of the limb that was treated.
  A minor amputation will be defined as below-the-ankle; and a major amputation will be defined as limb loss at or proximal to the transtibial level. Major amputations will be specified as below-the-knee and above-the-knee amputations.
Time Frame: 0 to 30 days
Population: ITT population. Per-subject basis analysis. The number of participants analyzed includes subjects who had available follow up data at that time frame.
Measure: Count of Participants; unit: Participants
Arm/Group | ESPRIT BVS
Number analyzed (Participants) | 35
Participants | 35

15. Secondary Outcome: Number of Participants With Limb Salvage (Freedom From Ipsilateral Major Amputations) of the Target Extremity
Description: as for outcome 14
Time Frame: 0 to 180 days
Population: as for outcome 14
Measure: Count of Participants; unit: Participants
Arm/Group | ESPRIT BVS
Number analyzed (Participants) | 35
Participants | 34

16. Secondary Outcome: Number of Participants With Limb Salvage (Freedom From Ipsilateral Major Amputations) of the Target Extremity
Description: as for outcome 14
Time Frame: 0 to 365 days
Population: as for outcome 14
Measure: Count of Participants; unit: Participants
Arm/Group | ESPRIT BVS
Number analyzed (Participants) | 35
Participants | 34

17. Secondary Outcome: Number of Participants With Limb Salvage (Freedom From Ipsilateral Major Amputations) of the Target Extremity
Description: as for outcome 14
Time Frame: 0 to 730 days
Population: as for outcome 14
Measure: Count of Participants; unit: Participants
Arm/Group | ESPRIT BVS
Number analyzed (Participants) | 35
Participants | 34

18. Secondary Outcome: Number of Participants With Limb Salvage (Freedom From Ipsilateral Major Amputations) of the Target Extremity
Description: as for outcome 14
Time Frame: 0 to 1095 days
Population: as for outcome 14
Measure: Count of Participants; unit: Participants
Arm/Group | ESPRIT BVS
Number analyzed (Participants) | 35
Participants | 30

19. Secondary Outcome: Number of Participants With Scaffold Thrombosis
Description: Scaffold Thrombosis is defined as total occlusion identified within the scaffold by arteriography and/or ultrasound that occurs within 30 days post- index procedure.
Time Frame: 0 to 1 month
Population: as for outcome 14
Measure: Count of Participants; unit: Participants
Arm/Group | ESPRIT BVS
Number analyzed (Participants) | 35
Participants | 0

20. Secondary Outcome: Scaffold Occlusion
Description: Number of participants with Scaffold Occlusion is defined as total occlusion identified within the scaffold by arteriography and/or ultrasound that occurs > 30 days post-index procedure.
Time Frame: 1 month
Population: as for outcome 14
Measure: Count of Participants; unit: Participants
Arm/Group | ESPRIT BVS
Number analyzed (Participants) | 35
Participants | 0

21. Secondary Outcome: Number of Participants With Scaffold Occlusion
Description: as for outcome 19
Time Frame: 6 months
Population: as for outcome 10
Measure: Count of Participants; unit: Participants
Arm/Group | ESPRIT BVS
Number analyzed (Participants) | 34
Participants | 0

22. Secondary Outcome: Number of Participants With Scaffold Occlusion
Description: Scaffold Occlusion is defined as total occlusion identified within the scaffold by arteriography and/or ultrasound that occurs > 30 days post-index procedure.
Time Frame: 1 year
Population: as for outcome 10
Measure: Count of Participants; unit: Participants
Arm/Group | ESPRIT BVS
Number analyzed (Participants) | 34
Participants | 1

23. Secondary Outcome: Number of Participants With Scaffold Occlusion
Description: as for outcome 22
Time Frame: 2 years
Population: as for outcome 10
Measure: Count of Participants; unit: Participants
Arm/Group | ESPRIT BVS
Number analyzed (Participants) | 33
Participants | 1

24. Secondary Outcome: Number of Participants With Scaffold Occlusion
Description: as for outcome 22
Time Frame: 0 to 3 years
Population: as for outcome 10
Measure: Count of Participants; unit: Participants
Arm/Group | ESPRIT BVS
Number analyzed (Participants) | 29
Participants | 1

25. Secondary Outcome: Number of Participants With Target Lesion Revascularization (TLR)
Description: Target lesion revascularization (TLR) is defined as any repeat percutaneous intervention of the target lesion or bypass surgery of the target vessel performed for restenosis or other complication of the target lesion.
Time Frame: 1 month
Population: as for outcome 9
Measure: Count of Participants; unit: Participants
Arm/Group | ESPRIT BVS
Number analyzed (Participants) | 35
Participants | 0

26. Secondary Outcome: Number of Participants With Target Lesion Revascularization (TLR)
Description: as for outcome 25
Time Frame: 6 months
Population: as for outcome 10
Measure: Count of Participants; unit: Participants
Arm/Group | ESPRIT BVS
Number analyzed (Participants) | 34
Participants | 0

27. Secondary Outcome: Number of Participants With Target Lesion Revascularization (TLR)
Description: as for outcome 25
Time Frame: 1 year
Population: as for outcome 10
Measure: Count of Participants; unit: Participants
Arm/Group | ESPRIT BVS
Number analyzed (Participants) | 34
Participants | 3

28. Secondary Outcome: Number of Participants With Target Lesion Revascularization (TLR)
Description: as for outcome 25
Time Frame: 2 years
Population: as for outcome 10
Measure: Count of Participants; unit: Participants
Arm/Group | ESPRIT BVS
Number analyzed (Participants) | 33
Participants | 4

29. Secondary Outcome: Number of Participants With Target Lesion Revascularization (TLR)
Description: as for outcome 25
Time Frame: 3 years
Population: as for outcome 10
Measure: Count of Participants; unit: Participants
Arm/Group | ESPRIT BVS
Number analyzed (Participants) | 29
Participants | 4

30. Secondary Outcome: Number of Participants With Ischemia-driven Target Lesion Revascularization (ID-TLR)
Description: A revascularization of the target lesion is considered ischemia driven if angiography shows a percent diameter stenosis ≥ 50% and there is worsening of the Rutherford Becker Clinical Category that is clearly referable to the target lesion. (worsening is defined as a deterioration (an increase) in the Rutherford Becker Clinical Category by more than 2 categories from the earliest post-procedural measurement or to a category 6.) An independent angiographic core laboratory should verify that the severity of percent diameter stenosis meets requirements for clinical indication and will overrule in cases where investigator reports are not in agreement.
Time Frame: 1 month
Population: as for outcome 9
Measure: Count of Participants; unit: Participants
Arm/Group | ESPRIT BVS
Number analyzed (Participants) | 35
Participants | 0

31. Secondary Outcome: Number of Participants With Ischemia-driven Target Lesion Revascularization (ID-TLR)
Description: as for outcome 30
Time Frame: 6 months
Population: as for outcome 10
Measure: Count of Participants; unit: Participants
Arm/Group | ESPRIT BVS
Number analyzed (Participants) | 34
Participants | 0

32. Secondary Outcome: Number of Participants With Ischemia-driven Target Lesion Revascularization (ID-TLR)
Description: as for outcome 30
Time Frame: 1 year
Population: as for outcome 10
Measure: Count of Participants; unit: Participants
Arm/Group | ESPRIT BVS
Number analyzed (Participants) | 34
Participants | 2

33. Secondary Outcome: Number of Participants With Ischemia-driven Target Lesion Revascularization (ID-TLR)
Description: as for outcome 30
Time Frame: 2 years
Population: as for outcome 10
Measure: Count of Participants; unit: Participants
Arm/Group | ESPRIT BVS
Number analyzed (Participants) | 33
Participants | 3

34. Secondary Outcome: Number of Participants With Ischemia-driven Target Lesion Revascularization (ID-TLR)
Description: as for outcome 30
Time Frame: 3 years
Population: as for outcome 10
Measure: Count of Participants; unit: Participants
Arm/Group | ESPRIT BVS
Number analyzed (Participants) | 29
Participants | 3

35. Secondary Outcome: Number of Participants With Ipsilateral Extremity Revascularization (IER)
Description: Ipsilateral extremity revascularization (IER) also called as Target extremity revascularization (TER). References to "target" lesion or extremity revised to "ipsilateral" lesion or extremity.
  Ipsilateral extremity revascularization (IER) is defined as any percutaneous intervention or surgical bypass of any segment of the ipsilateral extremity. The ipsilateral extremity is defined as the ipsilateral limb arteries proximal and distal to the target lesion, which includes upstream and downstream branches and excludes the target lesion itself.
Time Frame: 1 month
Population: as for outcome 9
Measure: Count of Participants; unit: Participants
Arm/Group | ESPRIT BVS
Number analyzed (Participants) | 35
Participants | 0

36. Secondary Outcome: Number of Participants With Ipsilateral Extremity Revascularization (IER)
Description: as for outcome 35
Time Frame: 6 months
Population: as for outcome 10
Measure: Count of Participants; unit: Participants
Arm/Group | ESPRIT BVS
Number analyzed (Participants) | 34
Participants | 0

37. Secondary Outcome: Number of Participants With Ipsilateral Extremity Revascularization (IER)
Description: as for outcome 35
Time Frame: 1 year
Population: as for outcome 10
Measure: Count of Participants; unit: Participants
Arm/Group | ESPRIT BVS
Number analyzed (Participants) | 34
Participants | 2

38. Secondary Outcome: Number of Participants With Ipsilateral Extremity Revascularization (IER)
Description: as for outcome 35
Time Frame: 2 years
Population: as for outcome 10
Measure: Count of Participants; unit: Participants
Arm/Group | ESPRIT BVS
Number analyzed (Participants) | 33
Participants | 3

39. Secondary Outcome: Number of Participants With Ipsilateral Extremity Revascularization (IER)
Description: as for outcome 35
Time Frame: 3 years
Population: as for outcome 10
Measure: Count of Participants; unit: Participants
Arm/Group | ESPRIT BVS
Number analyzed (Participants) | 29
Participants | 3

40. Secondary Outcome: Number of Participants With Primary Patency
Description: At the designated follow-up, intervention-free patency (< 50% diameter stenosis) since the initial procedure. Primary patency ends at the first occurrence of one of the following: reintervention for the purpose of treating the target lesion, total occlusion of the target lesion, surgical bypass of the target lesion, or amputation of the extremity due to target lesion restenosis or occlusion.
Time Frame: 1 month
Population: as for outcome 9
Measure: Count of Participants; unit: Participants
Arm/Group | ESPRIT BVS
Number analyzed (Participants) | 35
Participants | 0

41. Secondary Outcome: Number of Participants With Primary Patency
Description: as for outcome 40
Time Frame: 6 months
Population: as for outcome 10
Measure: Count of Participants; unit: Participants
Arm/Group | ESPRIT BVS
Number analyzed (Participants) | 34
Participants | 0

42. Secondary Outcome: Number of Participants With Primary Patency
Description: as for outcome 40
Time Frame: 1 year
Population: as for outcome 10
Measure: Count of Participants; unit: Participants
Arm/Group | ESPRIT BVS
Number analyzed (Participants) | 34
Participants | 7

43. Secondary Outcome: Number of Participants With Primary Patency
Description: as for outcome 40
Time Frame: 2 years
Population: as for outcome 10
Measure: Count of Participants; unit: Participants
Arm/Group | ESPRIT BVS
Number analyzed (Participants) | 33
Participants | 8

44. Secondary Outcome: Number of Participants With Primary Patency
Description: as for outcome 40
Time Frame: 3 years
Population: as for outcome 10
Measure: Count of Participants; unit: Participants
Arm/Group | ESPRIT BVS
Number analyzed (Participants) | 29
Participants | 9

45. Secondary Outcome: Number of Participants With Rutherford Becker Clinical Category Summary for the Treated Limb
Description: The Rutherford Becker clinical category is a scale to measure chronic limb ischemia.
  Category and Clinical Description:
  0 = Asymptomatic, no hemodynamically significant occlusive disease, 1 = Mild claudication, 2 = Moderate claudication, 3 = Severe claudication, 4 = Ischemic rest pain, 5 = Minor tissue loss, non-healing ulcer, or focal gangrene with diffuse pedal ischemia, 6 = Major tissue loss, extending above transmetatarsal level, functional foot no longer salvageable
Time Frame: 1 month
Population: as for outcome 10
Measure: Count of Participants; unit: Participants
Arm/Group | ESPRIT BVS
Number analyzed (Participants) | 33
Participants
  Category 0 | 28
  Category 1 | 4
  Category 2 | 1
  Category 3 | 0
  Category 4 | 0
  Category 5 | 0
  Category 6 | 0

46. Secondary Outcome: Number of Participants With Rutherford Becker Clinical Category Summary for the Treated Limb
Description: as for outcome 45
Time Frame: 6 months
Population: as for outcome 10
Measure: Count of Participants; unit: Participants
Arm/Group | ESPRIT BVS
Number analyzed (Participants) | 34
Participants
  Category 0 | 23
  Category 1 | 8
  Category 2 | 3
  Category 3 | 0
  Category 4 | 0
  Category 5 | 0
  Category 6 | 0

47. Secondary Outcome: Number of Participants With Rutherford Becker Clinical Category Summary for the Treated Limb
Description: as for outcome 45
Time Frame: 1 year
Population: as for outcome 10
Measure: Count of Participants; unit: Participants
Arm/Group | ESPRIT BVS
Number analyzed (Participants) | 34
Participants
  Category 0 | 25
  Category 1 | 4
  Category 2 | 3
  Category 3 | 2
  Category 4 | 0
  Category 5 | 0
  Category 6 | 0

48. Secondary Outcome: Number of Participants With Rutherford Becker Clinical Category Summary for the Treated Limb
Description: as for outcome 45
Time Frame: 2 years
Population: as for outcome 10
Measure: Count of Participants; unit: Participants
Arm/Group | ESPRIT BVS
Number analyzed (Participants) | 31
Participants
  Category 0 | 22
  Category 1 | 3
  Category 2 | 4
  Category 3 | 2
  Category 4 | 0
  Category 5 | 0
  Category 6 | 0

49. Secondary Outcome: Number of Participants With Rutherford Becker Clinical Category Summary for the Treated Limb
Description: as for outcome 45
Time Frame: 3 years
Population: as for outcome 10
Measure: Count of Participants; unit: Participants
Arm/Group | ESPRIT BVS
Number analyzed (Participants) | 25
Participants
  Category 0 | 19
  Category 1 | 3
  Category 2 | 3
  Category 3 | 0
  Category 4 | 0
  Category 5 | 0
  Category 6 | 0

50. Secondary Outcome: Ankle Brachial Index (ABI) for the Treated Limb
Description: The ABI is the ratio of the ankle to arm pressure, and it is calculated by dividing the systolic blood pressure in the ankle of the one leg by the higher of the two systolic blood pressures in the arms.
  An ABI of 0.9 - 1.3 is a normal range. A reduced ABI (less than 0.9) is consistent with peripheral artery occlusive disease, with values below 0.8 indicating moderate disease and below 0.5 indicates severe disease. A value greater than 1.3 is considered abnormal suggesting calcification of the walls of the arteries and noncompressible vessels, reflecting severe peripheral vascular disease. Subjects with ABI values greater than 1.3 will be excluded from the analysis.
  Calculation of the Ankle Brachial Index:
  (Highest Ankle Systolic Pressure/Highest Brachial Systolic Pressure = ABI)
Time Frame: At 1 month
Population: ITT population. Subjects with ABI values greater than 1.3 will be excluded from the analysis.
Measure: Mean (Standard Deviation); unit: ratio
Arm/Group | ESPRIT BVS
Number analyzed (Participants) | 30
ratio | 1.00 (0.11)

51. Secondary Outcome: Ankle Brachial Index (ABI) for the Treated Limb
Description: as for outcome 50
Time Frame: At 6 months
Population: ITT population. Subjects with ABI values greater than 1.3 will be excluded from the analysis.
Measure: Mean (Standard Deviation); unit: ratio
Arm/Group | ESPRIT BVS
Number analyzed (Participants) | 33
ratio | 0.99 (0.13)

52. Secondary Outcome: Ankle Brachial Index (ABI) for the Treated Limb
Description: as for outcome 50
Time Frame: At 1 year
Population: ITT population. Subjects with ABI values greater than 1.3 will be excluded from the analysis.
Measure: Mean (Standard Deviation); unit: ratio
Arm/Group | ESPRIT BVS
Number analyzed (Participants) | 34
ratio | 0.98 (0.15)

53. Secondary Outcome: Ankle Brachial Index (ABI) for the Treated Limb
Description: as for outcome 50
Time Frame: At 2 years
Population: ITT population. Subjects with ABI values greater than 1.3 will be excluded from the analysis.
Measure: Mean (Standard Deviation); unit: ratio
Arm/Group | ESPRIT BVS
Number analyzed (Participants) | 29
ratio | 0.96 (0.16)

54. Secondary Outcome: Ankle Brachial Index (ABI) for the Treated Limb
Description: as for outcome 50
Time Frame: At 3 years
Population: ITT population. Subjects with ABI values greater than 1.3 will be excluded from the analysis.
Measure: Mean (Standard Deviation); unit: ratio
Arm/Group | ESPRIT BVS
Number analyzed (Participants) | 23
ratio | 0.95 (0.13)

55. Secondary Outcome: Walking Impairment Questionnaire (WIQ) Scores
Description: Measured by the Walking Impairment Questionnaire (WIQ), a disease-specific instrument utilized to characterize walking ability through a questionnaire as an alternative to treadmill testing. It is a measure of subject-perceived walking performance for subjects with Peripheral Artery Disease (PAD) and/or intermittent claudication.
  The WIQ quantifies patient-reported walking speed, walking distance, and stair-climbing ability, respectively, on a scale of 0 (= worst) to 100 (= best).
Time Frame: At 1 month
Population: ITT population.The number of participants analyzed includes the subjects with available follow-up data at that time-point.The highest possible score for each domain is 100%, which indicates no difficulty. Lowest possible score for each domain is 0%, which indicates inability to perform the activity.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | ESPRIT BVS
Number analyzed (Participants) | 33
score on a scale
  Walking Distance Score | 86.02 (24.58)
  Walking Speed Score | 56.55 (21.99)
  Stair Climbing Score | 84.22 (23.93)

56. Secondary Outcome: Walking Impairment Questionaire Scores
Description: as for outcome 55
Time Frame: At 6 months
Population: ITT population.The number of participants analyzed includes the subjects with available follow-up data at that time-point. The highest score for each domain is 100%, which indicates no difficulty.Lowest possible score for each domain is 0%, which indicates inability to perform the activity.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | ESPRIT BVS
Number analyzed (Participants) | 34
score on a scale
  Walking Distance Score | 85.81 (24.66)
  Walking Speed Score | 52.79 (20.27)
  Stair Climbing Score | 81.25 (25.17)

57. Secondary Outcome: Walking Impairment Questionaire Scores
Description: as for outcome 55
Time Frame: At 1 year
Population: as for outcome 56
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | ESPRIT BVS
Number analyzed (Participants) | 34
score on a scale
  Walking Distance Score | 84.48 (29.86)
  Walking Speed Score | 52.69 (22.18)
  Stair Climbing Score | 87.50 (20.72)

58. Secondary Outcome: Walking Impairment Questionaire Scores
Description: as for outcome 55
Time Frame: At 2 years
Population: as for outcome 56
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | ESPRIT BVS
Number analyzed (Participants) | 31
score on a scale
  Walking Distance Score | 84.15 (25.70)
  Walking Speed Score | 50.93 (23.25)
  Stair Climbing Score | 83.60 (21.86)

59. Secondary Outcome: Walking Impairment Questionaire Scores
Description: as for outcome 55
Time Frame: At 3 years
Population: as for outcome 56
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | ESPRIT BVS
Number analyzed (Participants) | 25
score on a scale
  Walking Distance Score | 76.11 (25.86)
  Walking Speed Score | 56.74 (23.35)
  Stair Climbing Score | 75.50 (22.54)

60. Secondary Outcome: In-scaffold Peak Systolic Velocity (PSV)
Description: In-scaffold Peak Systolic Velocity (PSV) as Measured by Duplex Ultrasound
Time Frame: 1 month
Population: PSV was excluded from the analysis for subjects who had TLR prior to the duplex ultrasound and duplex ultrasound was not readable.
Measure: Mean (Standard Deviation); unit: cm/sec
Arm/Group | ESPRIT BVS
Number analyzed (Participants) | 29
cm/sec | 154.6 (46.8)

61. Secondary Outcome: In-scaffold Peak Systolic Velocity (PSV)
Description: In-scaffold Peak Systolic Velocity (PSV) as Measured by Duplex Ultrasound
Time Frame: 6 months
Population: as for outcome 60
Measure: Mean (Standard Deviation); unit: cm/sec
Arm/Group | ESPRIT BVS
Number analyzed (Participants) | 30
cm/sec | 151.5 (37.7)

62. Secondary Outcome: In-scaffold Peak Systolic Velocity (PSV)
Description: In-scaffold Peak Systolic Velocity (PSV) as Measured by Duplex Ultrasound
Time Frame: 1 year
Population: as for outcome 60
Measure: Mean (Standard Deviation); unit: cm/sec
Arm/Group | ESPRIT BVS
Number analyzed (Participants) | 30
cm/sec | 161.5 (72.6)

63. Secondary Outcome: In-scaffold Peak Systolic Velocity (PSV)
Description: In-scaffold Peak Systolic Velocity (PSV) as Measured by Duplex Ultrasound
Time Frame: 2 years
Population: as for outcome 60
Measure: Mean (Standard Deviation); unit: cm/sec
Arm/Group | ESPRIT BVS
Number analyzed (Participants) | 26
cm/sec | 162.7 (47.9)

64. Secondary Outcome: In-scaffold Peak Systolic Velocity (PSV)
Description: In-scaffold Peak Systolic Velocity (PSV) as Measured by Duplex Ultrasound
Time Frame: 3 years
Population: as for outcome 60
Measure: Mean (Standard Deviation); unit: cm/sec
Arm/Group | ESPRIT BVS
Number analyzed (Participants) | 17
cm/sec | 172.5 (67.2)

65. Secondary Outcome: In-scaffold Peak Systolic Velocity Ratio (PSVR)
Description: In-scaffold Peak Systolic Velocity Ratio (PSVR) as measured by duplex ultrasound
Time Frame: 1 month
Population: PSVR is excluded from the analysis for subjects who had TLR prior to the duplex ultrasound and duplex ultrasound was not readable.
Measure: Mean (Standard Deviation); unit: ratio
Arm/Group | ESPRIT BVS
Number analyzed (Participants) | 29
ratio | 1.26 (0.30)

66. Secondary Outcome: In-scaffold Peak Systolic Velocity Ratio (PSVR)
Description: Peak Systolic Velocity Ratio (PSVR) as measured by duplex ultrasound
Time Frame: 6 months
Population: as for outcome 65
Measure: Mean (Standard Deviation); unit: ratio
Arm/Group | ESPRIT BVS
Number analyzed (Participants) | 30
ratio | 1.35 (0.39)

67. Secondary Outcome: In-scaffold Peak Systolic Velocity Ratio (PSVR)
Description: Peak Systolic Velocity Ratio (PSVR) as measured by duplex ultrasound
Time Frame: 1 year
Population: as for outcome 65
Measure: Mean (Standard Deviation); unit: ratio
Arm/Group | ESPRIT BVS
Number analyzed (Participants) | 29
ratio | 1.66 (1.16)

68. Secondary Outcome: In-Scaffold Peak Systolic Velocity Ratio (PSVR)
Description: Peak Systolic Velocity Ratio (PSVR) as measured by duplex ultrasound
Time Frame: 2 years
Population: as for outcome 65
Measure: Mean (Standard Deviation); unit: ratio
Arm/Group | ESPRIT BVS
Number analyzed (Participants) | 24
ratio | 1.56 (0.49)

69. Secondary Outcome: In-scaffold Peak Systolic Velocity Ratio (PSVR)
Description: Peak Systolic Velocity Ratio (PSVR) as measured by duplex ultrasound
Time Frame: 3 years
Population: as for outcome 65
Measure: Mean (Standard Deviation); unit: ratio
Arm/Group | ESPRIT BVS
Number analyzed (Participants) | 15
ratio | 1.66 (0.57)

70. Secondary Outcome: Treated Site Percent Diameter Stenosis (%DS)
Description: Percent diameter stenosis (%DS) value calculated as 100 * (1 - MLD/RVD) using the mean values from two orthogonal views (when possible) by QA.
  * Reference Vessel Diameter (RVD)
  * Minimum Luminal Diameter(MLD)
Time Frame: post-procedure
Measure: Mean (Standard Deviation); unit: Percent Diameter stenosis
Arm/Group | ESPRIT BVS
Number analyzed (Participants) | 35
Percent Diameter stenosis
  In-Scaffold | 9.21 (7.18)
  In-Segment | 14.01 (8.25)

71. Secondary Outcome: Treated Site Percent Diameter Stenosis (%DS)
Description: as for outcome 70
Time Frame: 12 months
Population: The number of participants analyzed includes subjects who had available follow up data at that time frame.
Measure: Mean (Standard Deviation); unit: percent diameter stenosis
Units Other Than Participants: Target lesions
Arm/Group | ESPRIT BVS
Number analyzed (Participants) | 28
Number analyzed (Target lesions) | 28
percent diameter stenosis
  In-Scaffold | 31.88 (26.06)
  In-Segment | 35.24 (23.69)

72. Secondary Outcome: Treated Site Late Loss
Description: Mean in-lesion Late Loss is calculated as: (MLD post-procedure - MLD follow-up).
  The average of two orthogonal views (when possible) of the narrowest point within the area of assessment - in lesion, treated site or treated segment. Minimum Lumen Vessel Diameter (MLD) is visually estimated during angiography by the Investigator; it is measured during qualitative comparative analysis (QCA) by the Angiographic Core Lab.
Time Frame: 12 months
Population: The analysis population included subjects who had available follow up data at that time frame.
Measure: Mean (Standard Deviation); unit: Millimeter
Arm/Group | ESPRIT BVS
Number analyzed (Participants) | 28
Millimeter
  In-Scaffold | 1.30 (1.53)
  In-Segment | 1.23 (1.54)

73. Secondary Outcome: Binary Restenosis (≥50% DS)
Description: Binary restenosis is defined as the presence of a hemodynamically significant stenosis ≥ 50% as determined by duplex ultrasound or quantitative angiography (QA).
  Scaffold Stenosis ≥ 50% by Duplex Ultrasound Only
  In-scaffold %DS ≥ 50% by Arteriogram Only
Time Frame: 1 year
Population: ITT Population. The analysis population included subjects who had available follow up data at that time frame.
Measure: Number; unit: percentage of participants
Arm/Group | ESPRIT BVS
Number analyzed (Participants) | 34
percentage of participants | 20.6

74. Secondary Outcome: Quality of Life Measures: Physical Functioning (PF) Summary
Description: The 12-Item Short Form Health Survey (SF-12) questionnaire was used to determine general Quality of Life (QOL) measurements.
  SF-12® Health Survey is validated measure using 12 questions to measure functional health and well-being from the patient's point of view. Scores on the scale are 0% (indicating poor perceived health status) to 100% (indicating excellent perceived health status) possible.
Time Frame: At 1 month
Population: ITT population, per subject analysis. The number of participants analyzed includes the subjects with available follow-up data at that time point.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | ESPRIT BVS
Number analyzed (Participants) | 33
score on a scale | 51.26 (7.42)

75. Secondary Outcome: Quality of Life Measures: Physical Functioning (PF) Summary
Description: as for outcome 74
Time Frame: At 6 months
Population: as for outcome 74
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | ESPRIT BVS
Number analyzed (Participants) | 34
score on a scale | 49.14 (9.00)

76. Secondary Outcome: Quality of Life Measures: Physical Functioning (PF) Summary
Description: as for outcome 74
Time Frame: At 1 year
Population: as for outcome 74
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | ESPRIT BVS
Number analyzed (Participants) | 34
score on a scale | 50.66 (8.38)

77. Secondary Outcome: Quality of Life Measures: Physical Functioning (PF) Summary
Description: as for outcome 74
Time Frame: At 2 years
Population: as for outcome 74
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | ESPRIT BVS
Number analyzed (Participants) | 31
score on a scale | 46.49 (10.89)

78. Secondary Outcome: Quality of Life Measures: Physical Functioning (PF) Summary
Description: as for outcome 74
Time Frame: At 3 years
Population: as for outcome 74
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | ESPRIT BVS
Number analyzed (Participants) | 25
score on a scale | 46.16 (11.09)

79. Secondary Outcome: Quality of Life Measures: Role Physical (RP) Summary
Description: as for outcome 74
Time Frame: At 1 month
Population: as for outcome 74
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | ESPRIT BVS
Number analyzed (Participants) | 33
score on a scale | 49.64 (9.13)

80. Secondary Outcome: Quality of Life Measures: Role Physical (RP) Summary
Description: as for outcome 74
Time Frame: At 6 months
Population: as for outcome 74
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | ESPRIT BVS
Number analyzed (Participants) | 34
score on a scale | 50.27 (8.35)

81. Secondary Outcome: Quality of Life Measures: Role Physical (RP) Summary
Description: as for outcome 74
Time Frame: At 1 year
Population: as for outcome 74
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | ESPRIT BVS
Number analyzed (Participants) | 34
score on a scale | 49.72 (8.41)

82. Secondary Outcome: Quality of Life Measures: Role Physical (RP) Summary
Description: as for outcome 74
Time Frame: At 2 years
Population: as for outcome 74
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | ESPRIT BVS
Number analyzed (Participants) | 31
score on a scale | 47.37 (11.39)

83. Secondary Outcome: Quality of Life Measures: Role Physical (RP) Summary
Description: as for outcome 74
Time Frame: At 3 years
Population: as for outcome 74
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | ESPRIT BVS
Number analyzed (Participants) | 25
score on a scale | 47.59 (9.85)

84. Secondary Outcome: Quality of Life Measures: Bodily Pain (BP) Summary
Description: as for outcome 74
Time Frame: At 1 month
Population: as for outcome 74
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | ESPRIT BVS
Number analyzed (Participants) | 33
score on a scale | 50.34 (10.34)

85. Secondary Outcome: Quality of Life Measures: Bodily Pain (BP) Summary
Description: as for outcome 74
Time Frame: At 6 months
Population: as for outcome 74
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | ESPRIT BVS
Number analyzed (Participants) | 34
score on a scale | 49.65 (10.66)

86. Secondary Outcome: Quality of Life Measures: Bodily Pain (BP) Summary
Description: as for outcome 74
Time Frame: At 1 year
Population: as for outcome 74
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | ESPRIT BVS
Number analyzed (Participants) | 34
score on a scale | 52.05 (8.78)

87. Secondary Outcome: Quality of Life Measures: Bodily Pain (BP) Summary
Description: as for outcome 74
Time Frame: At 2 years
Population: as for outcome 74
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | ESPRIT BVS
Number analyzed (Participants) | 31
score on a scale | 50.54 (11.59)

88. Secondary Outcome: Quality of Life Measures: Bodily Pain (BP) Summary
Description: as for outcome 74
Time Frame: At 3 years
Population: as for outcome 74
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | ESPRIT BVS
Number analyzed (Participants) | 25
score on a scale | 48.88 (10.48)

89. Secondary Outcome: Quality of Life Measures: General Health (GH) Summary
Description: as for outcome 74
Time Frame: At 1 month
Population: as for outcome 74
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | ESPRIT BVS
Number analyzed (Participants) | 33
score on a scale | 48.46 (7.65)

90. Secondary Outcome: Quality of Life Measures: General Health (GH) Summary
Description: as for outcome 74
Time Frame: At 6 months
Population: as for outcome 74
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | ESPRIT BVS
Number analyzed (Participants) | 34
score on a scale | 47.09 (9.65)

91. Secondary Outcome: Quality of Life Measures: General Health (GH) Summary
Description: as for outcome 74
Time Frame: At 1 year
Population: as for outcome 74
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | ESPRIT BVS
Number analyzed (Participants) | 34
score on a scale | 47.97 (8.61)

92. Secondary Outcome: Quality of Life Measures: General Health (GH) Summary
Description: as for outcome 74
Time Frame: At 2 years
Population: as for outcome 74
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | ESPRIT BVS
Number analyzed (Participants) | 31
score on a scale | 46.97 (9.98)

93. Secondary Outcome: Quality of Life Measures: General Health (GH) Summary
Description: as for outcome 74
Time Frame: At 3 years
Population: as for outcome 74
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | ESPRIT BVS
Number analyzed (Participants) | 25
score on a scale | 47.84 (9.60)

94. Secondary Outcome: Quality of Life Measures: Vitality (VT) Summary
Description: as for outcome 74
Time Frame: At 1 month
Population: as for outcome 74
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | ESPRIT BVS
Number analyzed (Participants) | 33
score on a scale | 55.68 (8.99)

95. Secondary Outcome: Quality of Life Measures: Vitality (VT) Summary
Description: as for outcome 74
Time Frame: At 6 months
Population: as for outcome 74
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | ESPRIT BVS
Number analyzed (Participants) | 34
score on a scale | 56.04 (10.65)

96. Secondary Outcome: Quality of Life Measures: Vitality (VT) Summary
Description: as for outcome 74
Time Frame: At 1 year
Population: as for outcome 74
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | ESPRIT BVS
Number analyzed (Participants) | 34
score on a scale | 57.81 (10.80)

97. Secondary Outcome: Quality of Life Measures: Vitality (VT) Summary
Description: as for outcome 74
Time Frame: At 2 years
Population: as for outcome 74
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | ESPRIT BVS
Number analyzed (Participants) | 31
score on a scale | 57.49 (9.89)

98. Secondary Outcome: Quality of Life Measures: Vitality (VT) Summary
Description: as for outcome 74
Time Frame: At 3 years
Population: as for outcome 74
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | ESPRIT BVS
Number analyzed (Participants) | 24
score on a scale | 55.72 (11.86)

99. Secondary Outcome: Quality of Life Measures: Social Functioning (SF) Summary
Description: as for outcome 74
Time Frame: At 1 month
Population: as for outcome 74
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | ESPRIT BVS
Number analyzed (Participants) | 33
score on a scale | 53.51 (4.71)

100. Secondary Outcome: Quality of Life Measures: Social Functioning (SF) Summary
Description: as for outcome 74
Time Frame: At 6 months
Population: as for outcome 74
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | ESPRIT BVS
Number analyzed (Participants) | 34
score on a scale | 50.33 (9.95)

101. Secondary Outcome: Quality of Life Measures: Social Functioning (SF) Summary
Description: as for outcome 74
Time Frame: At 1 year
Population: as for outcome 74
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | ESPRIT BVS
Number analyzed (Participants) | 34
score on a scale | 52.71 (8.62)

102. Secondary Outcome: Quality of Life Measures: Social Functioning (SF) Summary
Description: as for outcome 74
Time Frame: At 2 years
Population: as for outcome 74
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | ESPRIT BVS
Number analyzed (Participants) | 31
score on a scale | 50.05 (12.10)

103. Secondary Outcome: Quality of Life Measures: Social Functioning (SF) Summary
Description: as for outcome 74
Time Frame: At 3 years
Population: as for outcome 74
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | ESPRIT BVS
Number analyzed (Participants) | 25
score on a scale | 50.11 (8.69)

104. Secondary Outcome: Quality of Life Measures: Role Emotional (RE) Summary
Description: as for outcome 74
Time Frame: At 1 month
Population: as for outcome 74
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | ESPRIT BVS
Number analyzed (Participants) | 33
score on a scale | 49.98 (9.42)

105. Secondary Outcome: Quality of Life Measures: Role Emotional (RE) Summary
Description: as for outcome 74
Time Frame: At 6 months
Population: as for outcome 74
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | ESPRIT BVS
Number analyzed (Participants) | 34
score on a scale | 51.31 (9.25)

106. Secondary Outcome: Quality of Life Measures: Role Emotional (RE) Summary
Description: as for outcome 74
Time Frame: At 1 year
Population: as for outcome 74
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | ESPRIT BVS
Number analyzed (Participants) | 34
score on a scale | 50.98 (10.70)

107. Secondary Outcome: Quality of Life Measures: Role Emotional (RE) Summary
Description: as for outcome 74
Time Frame: At 2 years
Population: as for outcome 74
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | ESPRIT BVS
Number analyzed (Participants) | 31
score on a scale | 49.04 (11.99)

108. Secondary Outcome: Quality of Life Measures: Role Emotional (RE) Summary
Description: as for outcome 74
Time Frame: At 3 years
Population: as for outcome 74
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | ESPRIT BVS
Number analyzed (Participants) | 25
score on a scale | 46.24 (13.24)

109. Secondary Outcome: Quality of Life Measures: Mental Health (MH) Summary
Description: as for outcome 74
Time Frame: At 1 month
Population: as for outcome 74
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | ESPRIT BVS
Number analyzed (Participants) | 33
score on a scale | 57.52 (7.94)

110. Secondary Outcome: Quality of Life Measures: Mental Health (MH) Summary
Description: as for outcome 74
Time Frame: At 6 months
Population: as for outcome 74
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | ESPRIT BVS
Number analyzed (Participants) | 34
score on a scale | 55.76 (9.98)

111. Secondary Outcome: Quality of Life Measures: Mental Health (MH) Summary
Description: as for outcome 74
Time Frame: At 1 year
Population: as for outcome 74
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | ESPRIT BVS
Number analyzed (Participants) | 34
score on a scale | 58.09 (10.39)

112. Secondary Outcome: Quality of Life Measures: Mental Health (MH) Summary
Description: as for outcome 74
Time Frame: At 2 years
Population: as for outcome 74
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | ESPRIT BVS
Number analyzed (Participants) | 31
score on a scale | 55.10 (10.54)

113. Secondary Outcome: Quality of Life Measures: Mental Health (MH) Summary
Description: as for outcome 74
Time Frame: At 3 years
Population: as for outcome 74
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | ESPRIT BVS
Number analyzed (Participants) | 24
score on a scale | 53.37 (11.60)

114. Secondary Outcome: Quality of Life Measures: Physical Component Summary (PCS)
Description: as for outcome 74
Time Frame: At 1 month
Population: as for outcome 74
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | ESPRIT BVS
Number analyzed (Participants) | 33
score on a scale | 48.61 (8.78)

115. Secondary Outcome: Quality of Life Measures: Physical Component Summary (PCS)
Description: as for outcome 74
Time Frame: At 6 months
Population: as for outcome 74
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | ESPRIT BVS
Number analyzed (Participants) | 34
score on a scale | 47.54 (9.53)

116. Secondary Outcome: Quality of Life Measures: Physical Component Summary (PCS)
Description: as for outcome 74
Time Frame: At 1 year
Population: as for outcome 74
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | ESPRIT BVS
Number analyzed (Participants) | 34
score on a scale | 48.56 (8.03)

117. Secondary Outcome: Quality of Life Measures: Physical Component Summary (PCS)
Description: as for outcome 74
Time Frame: At 2 years
Population: as for outcome 74
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | ESPRIT BVS
Number analyzed (Participants) | 31
score on a scale | 46.27 (11.13)

118. Secondary Outcome: Quality of Life Measures: Mental Component Summary (MCS)
Description: as for outcome 74
Time Frame: At 1 month
Population: as for outcome 74
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | ESPRIT BVS
Number analyzed (Participants) | 33
score on a scale | 55.67 (7.27)

119. Secondary Outcome: Quality of Life Measures: Physical Component Summary (PCS)
Description: as for outcome 74
Time Frame: At 3 years
Population: as for outcome 74
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | ESPRIT BVS
Number analyzed (Participants) | 25
score on a scale | 46.80 (11.00)

120. Secondary Outcome: Quality of Life Measures: Mental Component Summary (MCS)
Description: as for outcome 74
Time Frame: At 6 months
Population: as for outcome 74
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | ESPRIT BVS
Number analyzed (Participants) | 34
score on a scale | 55.12 (10.32)

121. Secondary Outcome: Quality of Life Measures: Mental Component Summary (MCS)
Description: as for outcome 74
Time Frame: At 1 year
Population: as for outcome 74
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | ESPRIT BVS
Number analyzed (Participants) | 34
score on a scale | 56.64 (11.33)

122. Secondary Outcome: Quality of Life Measures: Mental Component Summary (MCS)
Description: as for outcome 74
Time Frame: At 2 years
Population: as for outcome 74
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | ESPRIT BVS
Number analyzed (Participants) | 31
score on a scale | 54.97 (11.44)

123. Secondary Outcome: Quality of Life Measures: Mental Component Summary (MCS)
Description: as for outcome 74
Time Frame: At 3 years
Population: as for outcome 74
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | ESPRIT BVS
Number analyzed (Participants) | 25
score on a scale | 52.58 (11.69)

124. Secondary Outcome: Vascular Quality of Life (VascuQol) Scores Summary
Description: Vascular Quality of Life Questionnaire is defined as a disease specific quality of life (QOL) measure for subjects with chronic lower limb ischemia. Each item is rated as a seven point response scale, with a score of one being the worst and a score of seven the best possible. The total average score is the sum of all 25 items scores divided by 25. For each separate domain an average score can be calculated (sum of all items of one domain divided by the number of items of that domain). The highest score for each domain is 7, which indicates best health outcome.
  The domains include Activity Domain, Symptom Domain, Pain Domain, Emotional Domain, Social Domain.
Time Frame: At 1 month
Population: ITT population. The number of participants analyzed includes the subjects with available follow-up data at that time point.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | ESPRIT BVS
Number analyzed (Participants) | 33
score on a scale
  Activity Domain | 6.02 (0.90)
  Symptom Domain | 6.36 (0.60)
  Pain Domain | 6.26 (1.05)
  Emotional Domain | 6.35 (0.87)
  Social Domain | 6.44 (0.79)

125. Secondary Outcome: Vascular Quality of Life (VascuQol) Scores Summary
Description: as for outcome 124
Time Frame: At 6 months
Population: as for outcome 124
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | ESPRIT BVS
Number analyzed (Participants) | 34
score on a scale
  Activity Domain | 5.68 (0.98)
  Symptom Domain | 6.15 (0.91)
  Pain Domain | 6.20 (1.14)
  Emotional Domain | 6.31 (0.90)
  Social Domain | 6.40 (1.13)

126. Secondary Outcome: Vascular Quality of Life (VascuQol) Scores Summary
Description: as for outcome 124
Time Frame: At 1 year
Population: as for outcome 124
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | ESPRIT BVS
Number analyzed (Participants) | 34
score on a scale
  Activity Domain | 5.76 (0.83)
  Symptom Domain | 6.34 (0.91)
  Pain Domain | 6.21 (1.17)
  Emotional Domain | 6.44 (0.97)
  Social Domain | 6.68 (0.81)

127. Secondary Outcome: Vascular Quality of Life (VascuQol) Scores Summary
Description: as for outcome 124
Time Frame: At 2 years
Population: as for outcome 124
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | ESPRIT BVS
Number analyzed (Participants) | 31
score on a scale
  Activity Domain | 5.50 (1.05)
  Symptom Domain | 6.23 (0.82)
  Pain Domain | 6.02 (1.32)
  Emotional Domain | 6.22 (0.99)
  Social Domain | 6.42 (0.99)

128. Secondary Outcome: Vascular Quality of Life (VascuQol) Scores Summary
Description: as for outcome 124
Time Frame: At 3 years
Population: as for outcome 124
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | ESPRIT BVS
Number analyzed (Participants) | 24
score on a scale
  Activity Domain | 5.54 (0.90)
  Symptom Domain | 6.16 (0.90)
  Pain Domain | 5.69 (1.48)
  Emotional Domain | 6.10 (0.97)
  Social Domain | 6.21 (1.08)

ADVERSE EVENTS:
Time Frame: 3 years
Arm/Group | ESPRIT BVS
All-Cause Mortality (participants affected / at risk) | 0/35
Serious Adverse Events (participants affected / at risk) | 22/35
Other Adverse Events (participants affected / at risk) | 25/35
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | ESPRIT BVS (N=35)
Anemia (Blood and lymphatic system disorders) | 1
Bleeding (Blood and lymphatic system disorders) | 1
Hematuria (Blood and lymphatic system disorders) | 1
Acute Coronary Syndrome (Cardiac disorders) | 1
Angina (Cardiac disorders) | 2
Arrhythmia (Includes Brady And Tachy) (Cardiac disorders) | 1
Cerebrovascular accident (CVA) (Cardiac disorders) | 1
Coronary artery disease (CAD) - Coronary stenosis (Cardiac disorders) | 1
Dyspnea (Cardiac disorders) | 1
Myocardial Infarction - Unknown (Cardiac disorders) | 1
Other (Gastrointestinal disorders) | 3
Bronchitis (Infections and infestations) | 1
Other (Infections and infestations) | 1
Pneumonia (Infections and infestations) | 1
Urinary Tract Infection (Infections and infestations) | 1
Dissection (Injury, poisoning and procedural complications) | 1
Back Pain (Musculoskeletal and connective tissue disorders) | 2
Joint pain (Musculoskeletal and connective tissue disorders) | 2
Other (Musculoskeletal and connective tissue disorders) | 3
Stenosis (Musculoskeletal and connective tissue disorders) | 1
Trauma (Musculoskeletal and connective tissue disorders) | 2
Benign (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3
Flank Pain (Renal and urinary disorders) | 1
Renal Insufficiency (Renal and urinary disorders) | 1
Airway Obstruction (Respiratory, thoracic and mediastinal disorders) | 1
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1
Claudication (Vascular disorders) | 3
Ischemia (Vascular disorders) | 2
Occlusion (Vascular disorders) | 3
Peripheral artery disease (PAD) (Vascular disorders) | 1
Peripheral vascular disease (PVD) (Vascular disorders) | 2
Restenosis (Vascular disorders) | 2
Stenosis (Vascular disorders) | 5
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | ESPRIT BVS (N=35)
Anemia (Blood and lymphatic system disorders) | 2
Malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4
Angina (Cardiac disorders) | 3
Arrhythmia (Includes Brady And Tachy) (Cardiac disorders) | 2
Constipation (Gastrointestinal disorders) | 2
Other (Gastrointestinal disorders) | 3
Renal Insufficiency (Renal and urinary disorders) | 2
Pneumonia (Infections and infestations) | 2
Urinary Tract Infection (Infections and infestations) | 2
Pain (General disorders) | 2
Arthritis (Musculoskeletal and connective tissue disorders) | 2
Back Pain (Musculoskeletal and connective tissue disorders) | 3
Joint pain (Musculoskeletal and connective tissue disorders) | 3
Other (Musculoskeletal and connective tissue disorders) | 6
Trauma (Musculoskeletal and connective tissue disorders) | 3
Neuropathy (Nervous system disorders) | 2 — Neurologic Other Than Stroke
Hematoma (Injury, poisoning and procedural complications) | 2
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 3
Claudication (Vascular disorders) | 3
Ischemia (Vascular disorders) | 4
Occlusion (Vascular disorders) | 3
Peripheral vascular disease (PVD) (Vascular disorders) | 2
Restenosis (Vascular disorders) | 2
Stenosis (Vascular disorders) | 5
Bleeding (General disorders) | 1
Epistaxis (General disorders) | 1
Hematuria (Renal and urinary disorders) | 1
Benign cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Acute Coronary Syndrome (Cardiac disorders) | 1
CAD - Coronary stenosis (Cardiac disorders) | 1
Coronary Artery Disease (Cardiac disorders) | 1
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1
Myocardial Infarction - Unknown (Cardiac disorders) | 1
Cardiac/Hemodynamic : Other (Cardiac disorders) | 1
Structural Heart (Cardiac disorders) | 1
Thrombosis (Cardiac disorders) | 1
Bilary/Liver Disorder (Gastrointestinal disorders) | 1
Dysphagia (Gastrointestinal disorders) | 1
Gallstones (Gastrointestinal disorders) | 1
Bronchitis (Infections and infestations) | 1
Infection : Other (Infections and infestations) | 1
Viral, Bacterial And Fungal Infections (Infections and infestations) | 1
Abnormal Lab Test (Metabolism and nutrition disorders) | 1
Metabolic : Other (Metabolism and nutrition disorders) | 1
Depression (Psychiatric disorders) | 1
General disorders : Other (General disorders) | 1
Stenosis (Musculoskeletal and connective tissue disorders) | 1
Wound Complication Or Wound Infection (Musculoskeletal and connective tissue disorders) | 1
Epilepsy (Nervous system disorders) | 1
Neurologic Other Than Stroke: Other (Nervous system disorders) | 1
Peripheral Neuropathy (Nervous system disorders) | 1
Dissection (Injury, poisoning and procedural complications) | 1
Airway Obstruction (Respiratory, thoracic and mediastinal disorders) | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 1
Sepsis (Respiratory, thoracic and mediastinal disorders) | 1
Sleep Disorder (General disorders) | 1
Cerebrovascular accident (CVA) (Nervous system disorders) | 1
Peripheral artery disease (PAD) (Vascular disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No